CLINICAL TRIAL: NCT03120624
Title: Phase I Trial of Intravenous Administration of Vesicular Stomatitis Virus Genetically Engineered to Express Thyroidal Sodium Iodide Symporter (NIS) and Human Interferon Beta (hIFNb), in Patients With Metastatic or Recurrent Endometrial Cancer
Brief Title: VSV-hIFNbeta-NIS With or Without Ruxolitinib Phosphate in Treating Stage IV or Recurrent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1562; NCI-2017-00615 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1562 (Other: Mayo Clinic); R01CA207240 (NIH); 15-007000 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Endometrial Carcinoma; Recurrent Endometrial Adenocarcinoma; Recurrent Endometrial Carcinoma; Recurrent Endometrial Clear Cell Adenocarcinoma; Recurrent Endometrial Endometrioid Adenocarcinoma; Recurrent Endometrial Mixed Cell Adenocarcinoma; Recurrent Endometrial Serous Adenocarcinoma; Recurrent Endometrial Undifferentiated Carcinoma; Recurrent Uterine Corpus Carcinosarcoma; Stage IV Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Biopsy; Magnetic Resonance Spectroscopy; sodium-iodide symporter; ruxolitinib; Sodium Pertechnetate Tc 99m; Radionuclide Generators; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (VSV-hIFNbeta-NIS, TFB-PET, biopsy) (Experimental): Patients receive VSV-hIFNbeta-NIS IV over 60-90 minutes on day 1. After 2 days, patients receive technetium Tc-99m sodium pertechnetate IV, and about 30 minutes later, receive fluorine F18 tetrafluoroborate IV and undergo TFB-PET imaging. If previous imaging data are positive, patients receive technetium Tc-99m sodium pertechnetate IV and fluorine F18 tetrafluoroborate IV and undergo another TFB-PET imaging between 7-10 days and on 15 days if needed after VSV-hIFNbeta-NIS infusion. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo CT throughout the study. Patients also undergo mouth rinse, buccal swab and urine on study and blood sample collection throughout the study. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo image-guided biopsy of accessible tumor on day 29.
  Interventions: Procedure: Biopsy; Procedure: Computed Tomography; Other: Fluorine F 18 Tetrafluoroborate; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Drug: Technetium Tc-99m Sodium Pertechnetate; Procedure: Biospecimen Collection
- Arm B (ruxolitinib, VSV-hIFNbeta-NIS, SPECT/CT,TFB-PET,biopsy) (Experimental): Patients receive ruxolitinib phosphate PO BID on days -3 to 9. Patients also receive VSV-hIFNbeta-NIS IV over 60-90 minutes on day 1. After 2 days, patients receive technetium Tc-99m sodium pertechnetate IV, and about 30 minutes later, receive fluorine F18 tetrafluoroborate IV and undergo TFB-PET imaging. If previous imaging data are positive, patients receive technetium Tc-99m sodium pertechnetate IV and undergo fluorine F18 tetrafluoroborate IV and undergo another TFB-PET imaging between 7-10 days and on 15 days if needed after VSV-hIFNbeta-NIS infusion. Patients also undergo CT throughout the study. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo image-guided biopsy of accessible tumor on day 29. Patients also undergo mouth rinse, buccal swab and urine on study and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Computed Tomography; Other: Fluorine F 18 Tetrafluoroborate; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Drug: Ruxolitinib Phosphate; Drug: Technetium Tc-99m Sodium Pertechnetate; Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biopsy — Undergo image-guided biopsy
  Other Names: Biopsy Type; BIOPSY_TYPE; Bx
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Fluorine F 18 Tetrafluoroborate — Given IV
  Other Names: 18F-Tetrafluoroborate; 18F-TFB
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Undergo TFB-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Biological: Recombinant Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter — Given IV
  Other Names: Oncolytic VSV-hIFNbeta-NIS; Vesicular Stomatitis Virus-expressing Human Interferon Beta and Sodium-Iodide Symporter; Voyager-V1; VSV-expressing hIFNb and NIS; VSV-hIFNb-NIS; VSV-hIFNbeta-NIS; VV1
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: 1092939-17-7; INCB-18424 Phosphate; Jakafi; Jakavi
  Arms: Arm B (ruxolitinib, VSV-hIFNbeta-NIS, SPECT/CT,TFB-PET,biopsy)
Drug: Technetium Tc-99m Sodium Pertechnetate — Given IV
  Other Names: Pertscan-99m; Sodium Pertechnetate (Na99mtco4); Tc 99m Generator; Ultra-Technekow FM
Procedure: Biospecimen Collection — Undergo mouth rinse, buccal swab, urine, and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I trial studies the side effects and best dose of vesicular stomatitis virus-human interferon beta-sodium iodide symporter (VSV-hIFNbeta-NIS) with or without ruxolitinib phosphate in treating patients with stage IV endometrial cancer or endometrial cancer that has come back. The study virus, VSV-hIFNbeta-NIS, has been changed so that it has restricted ability to spread to tumor cells and not to healthy cells. It also contains a gene for a protein, NIS, which helps the body concentrate iodine making it possible to track where the virus goes. VSV-hIFNbeta-NIS may be able to kill tumor cells without damaging normal cells. Ruxolitinib phosphate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving VSV-hIFNbeta-NIS with ruxolitinib phosphate may work better in treating patients with endometrial cancer compared to VSV-hIFNbeta-NIS alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the optimal dose schedule, safety and tolerability as measured by the incidence of significant toxicity of VSV-hIFNbeta-NIS in immunocompetent patients with metastatic and/or recurrent endometrial cancer (EC).

SECONDARY OBJECTIVES:

I. To determine the toxicity profile of VSV-hIFNbeta-NIS (alone and in combination with ruxolitinib phosphate [ruxolitinib]).

II. To determine the time course of viral gene expression and virus elimination, and the biodistribution of virally infected cells at various times points after infection with VSV-hIFNbeta-NIS (alone and in combination with ruxolitinib) using fluorine F18 tetrafluoroborate (TFB)-positron emission tomography (PET) imaging.

III. To assess virus replication, viremia; viral shedding in urine and respiratory secretions; and virus persistence after intravenous (IV) administration of VSV-hIFNbeta-NIS (alone and in combination with ruxolitinib).

IV. To monitor humoral responses to the injected virus. V. To estimate the tumor response rate and overall survival.

CORRELATIVE OBJECTIVES:

I. To determine the pharmacokinetic (PK) profile of VSV-IFNbeta-NIS in patients with EC by measurement of VSV-IFNbeta-NIS in blood by reverse transcriptase polymerase chain reaction (RT-PCR).

II. To characterize the pharmacodynamics (PD) of VSV-IFNbeta-NIS by way of measuring serum interferon-beta and also VSV-RT-PCR of VSV-IFNbeta-NIS listed above.

III. Assess CD8+ T cell (both general and VSV-IFNbeta-NIS specific) and natural killer (NK) cell responses.

IV. Gene expression analysis pre- and post-virotherapy. V. Evaluate transcription of interferon mediated genes (protein kinase R, the death receptor-TRAIL, 2'-5' oligoadenylate/RNAse L proteins, heat shock proteins [Hsp 60/70/90], major histocompatibility class antigens and IRF-7).

VI. Assess presence of VSV in tumor and normal tissues subsequent to administration of IV VSV-IFNbeta-NIS.

OUTLINE: This is a dose-escalation study of VSV-hIFNbeta-NIS. Patients are randomized to 1 of 2 arms.

ARM A (EFFECTIVE AS OF 1/10/2023, GROUP A IS PERMANENTLY CLOSED TO ACCRUAL): Patients receive VSV-hIFNbeta-NIS IV over 60-90 minutes on day 1. After 2 days, patients receive technetium Tc-99m sodium pertechnetate IV, and about 30 minutes later, receive fluorine F18 tetrafluoroborate IV and undergo TFB-PET imaging. If previous imaging data are positive, patients receive technetium Tc-99m sodium pertechnetate IV, fluorine F18 tetrafluoroborate IV and undergo another TFB-PET imaging between 7-10 days and on 15 days if needed after VSV-hIFNbeta-NIS infusion. Patients also undergo computed tomography (CT) throughout the study. Patients also undergo mouth rinse, buccal swab and urine on study and blood sample collection throughout the study. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo image-guided biopsy of accessible tumor on day 29.

ARM B: Patients receive ruxolitinib phosphate orally (PO) twice daily (BID) on days -3 to 9. Patients also receive VSV-hIFNbeta-NIS IV over 60-90 minutes on day 1. After 2 days, patients receive technetium Tc-99m sodium pertechnetate IV, and about 30 minutes later, receive fluorine F18 tetrafluoroborate IV and undergo TFB-PET imaging. If previous imaging data are positive, patients receive technetium Tc-99m sodium pertechnetate IV and fluorine F18 tetrafluoroborate IV and undergo another TFB-PET imaging between 7-10 days and on 15 days if needed after VSV-hIFNbeta-NIS infusion. Patients also undergo CT throughout the study. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo image-guided biopsy of accessible tumor on day 29. Patients also undergo mouth rinse, buccal swab and urine on study and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at day 29, every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Measurable stage IVA, stage IVB (with or without measurable disease) or recurrent (with or without measurable disease) endometrial carcinoma

  * NOTE: histologic confirmation of the original primary tumor is required; patients with the following histologic epithelial cell types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, carcinosarcoma, adenocarcinoma not otherwise specified (NOS)
  * NOTE: measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)
* Group A only: Largest tumor diameter =< 5 cm

  * NOTE: Group B patients have no maximum tumor size
* Absolute neutrophil count (ANC) >= 1500/uL (obtained =< 14 days prior to registration)
* Platelet count (PLT) >= 100,000/uL (obtained =< 14 days prior to registration)
* Hemoglobin >= 10 g/dL (obtained =< 14 days prior to registration)
* Creatinine =< 2.0 mg/dL (obtained =< 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)

  * NOTE: if baseline liver disease, Child Pugh score not exceeding class A
* Total bilirubin =< 1.5 x ULN (obtained =< 14 days prior to registration)
* International normalized ratio (INR)/prothrombin time (PT), activated partial thromboplastin time (aPTT) =< 1.4 x ULN (obtained =< 14 days prior to registration) unless on therapeutic warfarin then INR/PT =< 3.5
* Ability to provide written informed consent
* Willingness to return to Mayo Clinic in Rochester, Minnesota for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Willingness to provide mandatory biological specimens for research purposes
* Prior therapy:

  * Any number of prior chemotherapy regimens and/or targeted therapies and/or prior external beam radiation therapy and/or prior hormonal therapy for endometrial cancer are allowed provided the last treatment was >= 4 weeks prior to registration
  * Vaginal brachytherapy may have been administered at any time prior to registration

Exclusion Criteria:

* Availability of and patient acceptance of curative therapy
* Active infection requiring treatment, including any active viral infection, =< 5 days prior to registration
* Active or latent tuberculosis or hepatitis
* Known untreated or symptomatic brain metastases
* Any of the following prior therapies:

  * Chemotherapy < 4 weeks prior to registration
  * Targeted biologic therapy < 4 weeks prior to registration
  * Immunotherapy < 4 weeks prior to registration
  * Any viral or gene therapy prior to registration
  * External beam radiotherapy < 4 weeks prior to registration

    * NOTE: Vaginal brachytherapy may be performed at any time prior to registration
* New York Heart Association classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or uncontrolled current cardiac arrhythmias (atrial fibrillation or supraventricular tachycardia [SVT])
* Active central nervous system (CNS) disorder or seizure disorder or known CNS disease or neurologic symptomatology
* Human immunodeficiency virus (HIV) positive test result or other immunodeficiency or immunosuppression
* History of hepatitis B or C or chronic hepatitis
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (used for a non-Food and Drug Administration [FDA] approved indication and in the context of a research investigation)
* Treatment with oral/systemic corticosteroids, with the exception of topical or inhaled steroids
* Exposure to household contacts =< 15 months old or household contact with known immunodeficiency
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons or persons of reproductive ability who are unwilling to use effective contraception
  * Nursing persons
* Any other pathology or condition that the principal investigator deems to negatively impact treatment safety
* Any immunotherapy-related adverse events Common Terminology Criteria for Adverse Events (CTCAE) > grade 1 at the time of registration
* Receipt of a live virus vaccine =< 2 months prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2028-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie N. Bakkum-Gamez, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A Dose Level 1; Cohort A Dose Level 2; Cohort A Dose Level 3; Cohort A Dose Level 4: Patients receive VSV-hIFNbeta-NIS IV over 60-90 minutes on day 1. After 2 days, patients receive technetium Tc-99m sodium pertechnetate IV, and about 30 minutes later, receive fluorine F18 tetrafluoroborate IV and undergo TFB-PET imaging. If previous imaging data are positive, patients receive technetium Tc-99m sodium pertechnetate IV and fluorine F18 tetrafluoroborate IV and undergo another TFB-PET imaging between 7-10 days and on 15 days if needed after VSV-hIFNbeta-NIS infusion. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo CT throughout the study. Patients also undergo mouth rinse, buccal swab and urine on study and blood sample collection throughout the study. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo image-guided biopsy of accessible tumor on day 29.
- Cohort B Dose Level 1; Cohort B Dose Level 2; Cohort B Dose Level 3; Cohort B Dose Level 4: Patients receive ruxolitinib phosphate PO BID on days -3 to 9. Patients also receive VSV-hIFNbeta-NIS IV over 60-90 minutes on day 1. After 2 days, patients receive technetium Tc-99m sodium pertechnetate IV, and about 30 minutes later, receive fluorine F18 tetrafluoroborate IV and undergo TFB-PET imaging. If previous imaging data are positive, patients receive technetium Tc-99m sodium pertechnetate IV and undergo fluorine F18 tetrafluoroborate IV and undergo another TFB-PET imaging between 7-10 days and on 15 days if needed after VSV-hIFNbeta-NIS infusion. Patients also undergo CT throughout the study. Biopsy of accessible NIS image-positive tumors may occur after any imaging. Patients also undergo image-guided biopsy of accessible tumor on day 29. Patients also undergo mouth rinse, buccal swab and urine on study and blood sample collection throughout the study.
Period: Overall Study
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort A Dose Level 3 | Cohort A Dose Level 4 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Started | 3 | 10 | 3 | 6 | 3 | 3 | 3 | 3
Completed | 3 | 9 | 3 | 6 | 3 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only patients that started treatment are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort A Dose Level 3 | Cohort A Dose Level 4 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4 | Total
Number analyzed (Participants) | 3 | 9 | 3 | 6 | 3 | 3 | 3 | 3 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (8.14) | 65.6 (7) | 62.7 (5.03) | 60.2 (16.3) | 66 (11.53) | 68.3 (2.08) | 67 (2.65) | 63.7 (6.43) | 63.5 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 3 | 6 | 3 | 3 | 3 | 3 | 33
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 9 | 3 | 5 | 3 | 2 | 3 | 3 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 8 | 3 | 5 | 2 | 2 | 3 | 3 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: Graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4. DLT is defined as one of the following events deemed related to the study drug; Grade 2+ allergic reaction or cytokine release syndrome, or any grade 3+ with the exception of lymphopenia or other related events (e.g., anemia, white blood cell count decreased), which will not be considered a dose limiting toxicity. Grade ≥3 flu-like symptoms, fever, nausea, vomiting, dehydration, diarrhea, headache, myalgia, fatigue, ALT increased, or AST increased, will also not be considered as a dose limiting toxicity as they are anticipated toxicities of treatment.
Time Frame: 28 days
Population: All treated patients are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort A Dose Level 3 | Cohort A Dose Level 4 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 3 | 9 | 3 | 6 | 3 | 3 | 3 | 3
Participants | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0

2. Secondary Outcome: Incidence of Adverse Events
Description: Graded according to the NCI CTCAE version 4. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables. Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and related confidence intervals.
Time Frame: Up to 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Number of Clinical Responses
Description: Defined as complete response, partial response, or stable disease assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Will be summarized by simple descriptive summary statistics across all patients in each group as well as by dose level and primary type of cancer (EC).
Time Frame: Up to 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Viral Replication and Shedding in Blood, Throat Washings, Urine, and Buccal Swabs Assessed Via Quantitative Reverse Transcriptase Polymerase Chain Reaction
Description: Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations with other outcome measures will be carried out by standard parametric and non-parametric tests (e.g. Pearson's and Spearman's rho).
Time Frame: Up to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Count of Patients With Positive Virus Spread.
Description: Virus spread will be ssessed via single-photon emission computed tomography/computed tomography and will be correlated with tumor distribution.
Time Frame: 10 days
Population: Tomography was only conducted on patients accrued prior to 8/6/2021 due to all of the scans failing to observe any virus spread. The burden to patients and research resources was deemed unacceptable for no scientific benefit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort A Dose Level 3 | Cohort A Dose Level 4 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
Number analyzed (Participants) | 3 | 9 | 3 | 5 | 3 | 2 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Time Until Treatment Related Grade 3+ Toxicity
Description: Graded according to the NCI CTCAE version 4. Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and related confidence intervals. The effect of dose and ancillary dichotomized covariates such as age will be explored using logrank testing involving one covariate at a time.
Time Frame: Up to 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Time Until Hematologic Nadirs (White Blood Cells, Absolute Neutrophil Count, Platelets)
Description: Simple summary statistics will be supplemented with Kaplan-Meier survival estimates and related confidence intervals. The effect of dose and ancillary dichotomized covariates such as age will be explored using logrank testing involving one covariate at a time.
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 1 year and mortality was followed for 63 months.
Arm/Group | Cohort A Dose Level 1 | Cohort A Dose Level 2 | Cohort A Dose Level 3 | Cohort A Dose Level 4 | Cohort B Dose Level 1 | Cohort B Dose Level 2 | Cohort B Dose Level 3 | Cohort B Dose Level 4
All-Cause Mortality (participants affected / at risk) | 2/3 | 7/9 | 3/3 | 4/6 | 2/3 | 2/3 | 3/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/9 | 0/3 | 4/6 | 1/3 | 1/3 | 0/3 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 3/3 | 6/6 | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Dose Level 1 (N=3) | Cohort A Dose Level 2 (N=9) | Cohort A Dose Level 3 (N=3) | Cohort A Dose Level 4 (N=6) | Cohort B Dose Level 1 (N=3) | Cohort B Dose Level 2 (N=3) | Cohort B Dose Level 3 (N=3) | Cohort B Dose Level 4 (N=3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Dose Level 1 (N=3) | Cohort A Dose Level 2 (N=9) | Cohort A Dose Level 3 (N=3) | Cohort A Dose Level 4 (N=6) | Cohort B Dose Level 1 (N=3) | Cohort B Dose Level 2 (N=3) | Cohort B Dose Level 3 (N=3) | Cohort B Dose Level 4 (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 5 (26) | 3 (15) | 6 (33) | 3 (8) | 3 (20) | 3 (16) | 1 (8)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 2 (5) | 0 (0) | 1 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 3 (8) | 2 (5) | 3 (9) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (5) | 8 (27) | 2 (10) | 5 (23) | 3 (8) | 1 (2) | 1 (2) | 2 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (19) | 2 (2) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
Chills (General disorders) | 1 (2) | 7 (9) | 3 (4) | 5 (8) | 3 (6) | 0 (0) | 3 (3) | 3 (3)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (7) | 0 (0) | 1 (5)
Fatigue (General disorders) | 2 (12) | 8 (30) | 3 (22) | 5 (34) | 3 (24) | 2 (14) | 1 (8) | 2 (13)
Fever (General disorders) | 1 (7) | 9 (16) | 3 (4) | 3 (8) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (6) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Activated partial throm time prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (16) | 3 (6) | 5 (17) | 0 (0) | 2 (8) | 1 (3) | 1 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (16) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (4) | 2 (13)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 6 (18) | 3 (7) | 5 (22) | 1 (3) | 2 (9) | 2 (5) | 2 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 4 (11) | 1 (3) | 5 (25) | 2 (2) | 2 (8) | 1 (5) | 2 (8)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (5) | 9 (39) | 3 (19) | 6 (36) | 3 (8) | 3 (18) | 3 (7) | 3 (7)
Neutrophil count decreased (Investigations) | 2 (5) | 4 (10) | 1 (5) | 2 (7) | 2 (2) | 2 (7) | 2 (6) | 2 (4)
Platelet count decreased (Investigations) | 2 (9) | 7 (30) | 3 (13) | 5 (24) | 2 (9) | 2 (11) | 2 (6) | 2 (5)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (7) | 4 (19) | 1 (9) | 2 (5) | 1 (4) | 2 (10) | 2 (7) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 4 (9) | 1 (6) | 1 (5) | 2 (4) | 2 (6) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 3 (10) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 5 (17) | 3 (9) | 5 (15) | 2 (5) | 3 (13) | 3 (8) | 2 (11)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4) | 3 (7) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (3) | 1 (3)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (8) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 2 (8) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 3 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (10) | 3 (8) | 2 (8) | 2 (4) | 2 (5) | 2 (2) | 1 (5)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (6) | 1 (7) | 1 (3) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 6 (13) | 2 (5) | 6 (15) | 2 (5) | 2 (9) | 2 (7) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03120624/Prot_SAP_000.pdf